CLINICAL TRIAL: NCT04945187
Title: Systematic Nurse-Led Consultations Based on Electronic Patient-Reported Outcome Among Women With Gynecological Cancer During Chemotherapy (The CONNECT Study)
Brief Title: Patient-Reported Outcomes Among Women Wtih Gynecological Cancer (The CONNECT Study)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: The Novo Nordic Foundation (Other)
Responsible Party: Principal Investigator, Helle Pappot, Professor, Clinical Oncologist, Consultant, DMSc, Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: Copenhagen University Hospital
Record Dates: First submitted 2021-05-11; First posted 2021-06-30 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Gynecologic Cancer; Gynecologic Neoplasm; Ovarian Cancer; Endometrial Cancer
Keywords: Patient-reported outcome; Electronic patient-reported outcome; Nurse-led consultations; Quality of life
MeSH Terms: conditions — Genital Neoplasms, Female; Ovarian Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Intervention Model Description: A prospective, sequential cohort study with comparisons between non-equivalent groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (No Intervention): No intervention. This arm will continue standard clinical practice consisting of clinical assessment regarding side effects and management before each cycle of chemotherapy conducted by physicians.
- Intervention group (Experimental): Intervention: This arm will be assigned to the intervention which will be nurse-led consultations based on electronic patient-reported outcomes. The patients will report ePRO weekly during chemotherapy and the answers will be used proactively in the nurse-led consultations. Nurses will conduct the clinical assessment regarding side effects and management before each cycle of chemotherapy.
  Interventions: Other: Nurse-led consultations based on electronic patient-reported outcomes

INTERVENTIONS:
Other: Nurse-led consultations based on electronic patient-reported outcomes — The patients will weekly answer electronic patient-reported outcomes during chemotherapy and the answers will be used proactive in nurse-led consultations.
  Arms: Intervention group

SUMMARY:
Systematic nurse-led consultations based on electronic patient-reported outcomes (ePRO) will be tested among women with ovarian - and endometrial cancer receiving first-line chemotherapy.

DETAILED DESCRIPTION:
Women with ovarian- and endometrial cancer often experiences a high disease and treatment-related physical and psychological burden. Patient-reported outcomes (PRO) have the potential to improve patient-clinician communication, symptom management, involvement, and quality of life. Electronic patient-reported outcomes (ePRO) can facilitate appropriate and continuous symptom monitoring reported by the patients. Nurses are with their holistic approach and their specialized knowledge and experience in a prominent position to address and facilitate symptom-management in a multidisciplinary context.

The overall aim of this study is to develop a model of care for systematic nurse-led consultations based on ePRO facilitating symptom management and to investigate how these consultations can be a part of the multidisciplinary treatment regimen for women with ovarian- and endometrial cancer receiving chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 18 years
* Newly diagnosis of ovarian- or endometrial cancer
* Scheduled to receive first-line standard chemotherapy
* Having an active email, internet access and a device
* Able to understand, read and speak Danish

Exclusion Criteria:

* Severe cognitive impairments/psychiatric disorder
* Participating in other interventional clinical trials

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 130 (Estimated)
Dates: Start 2021-05-17 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Quality of life measured by EORTC QLQ C-30 until 9 months. | Change from baseline to 9 months.
  EORTC QLQ C-30, a higher score indicates better quality of life (range 0-100). Measured at four time-points.

SECONDARY OUTCOMES:
Change from baseline in disease-specific Quality of life using the EORTC QLQ-OV28 Ovarian Module until 9 months. | Change from baseline to 9 months.
  Includes 28 questions. Measured at four time-points.
Change from baseline in disease-specific Quality of life using the EORTC QLQ-EN24 Endometrial Module until 9 months. | 9 months; at baseline (0 months), 3, 6 and 9 months.
  Includes 24 questions. Measured at four time-points.
Change from baseline in Hospital Anxiety and Depression Scale (HADS) until 9 months. | Change from baseline to 9 months.
  Includes 14 questions, addressing anxiety and depressive symptoms with 7 items each in the previous 7 days. Measured at four time-points.
Change from baseline in Self-efficacy for managing chronic disease 6-item scale until 9 months. | Change from baseline to 9 months.
  A 6-item scale measuring patient's perceived self-efficacy on a 10 point Likert Scale. Measured at four time-points.
Common Terminology Criteria for Adverse Events (CTCAE), an objective grading of the patients symptoms. | Before each cycle of chemotherapy, in total 6 cycles. A cycle is 21 days.
  Scale 0-4, where 0 is no/nothing and 4 is severe.

CONTACTS AND LOCATIONS:
Overall Officials: Mille Christiansen, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No